CLINICAL TRIAL: NCT03115944
Title: A Multi-Center Pilot Study to Assess the Safety and Efficacy of the vShape Ultra UltraSpeed Handpiece for Abdomen Circumference Reduction
Brief Title: Pro00019086 - Ultra Circumference Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alma Lasers Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlmaLasersInc
Record Dates: First submitted 2016-10-13; First posted 2017-04-14 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-04

CONDITIONS: Circumference Reduction of Abdomen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UltraSpeed Treatment (Experimental): UltraSpeed ultrasound treatments
  Interventions: Device: Alma vShape Ultra

INTERVENTIONS:
Device: Alma vShape Ultra — UltraSpeed ultrasound treatment, a series of four treatments
  Other Names: UltraSpeed

SUMMARY:
A Multi-Center Pilot Study to Assess the Safety and Efficacy of the VShape Ultra UltraSpeed Handpiece for Abdomen Circumference Reduction

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* Female and male subjects, between 18 and 45 years of age at the time of enrollment.
* Fitzpatrick Skin Type I to VI.
* Fat thickness of at least 1.5 cm in the treated area (measured by calibrated caliper).
* BMI interval: BMI between 20 to 30 (normal to overweight, but not obese).
* If female, not pregnant or lactating, must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
* In addition, negative urine pregnancy test as tested before each treatment and at the last follow-up visit for women with childbearing potential (e.g., not menopausal).
* General good health confirmed by medical history and skin examination of the treated area.
* Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
* Willingness to refrain from a change in diet / exercise / medication regimen for the entire course of the study.
* Willing to have photographs and images taken of the treated areas to be used, de-identified in evaluations, publications and presentations.

Exclusion Criteria:

* History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker / defibrillator, abnormal aortic aneurism.
* Known hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease.
* Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
* Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
* Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone.
* Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction.
* Previous body contouring procedures in the treatment area within 12 months.
* History of skin disease in the treatment area; known tendency to form keloids or poor wound healing.
* Suffering from significant skin conditions in the treatment areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during treatment course.
* Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions), including depressed scars in the treatment area.
* Very poor skin quality (i.e., severe laxity).
* Abnormal wall diastasis or hernia on physical examination.
* Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months.
* Obesity (BMI above 30)
* Childbirth within the last 12 months or breastfeeding women.
* Any acute or chronic condition which, in the opinion of the Investigator may exclude the candidate / patient from entry into the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Average Circumference Reduction as Measured by Skin Fold and Photography | 4 Treatments over 4 Weeks
  Skin fold measure utilizes caliper and photography utilizes Galaxy medical camera with extrapolation of measuring dot. Last measurement taken 14 days after final treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AboutSkin Dermatology, Greenwood Village, Colorado
  - Maryland Plastic Surgery, Glen Burnie, Maryland
  - Dr. Brian S. Biesman, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided